CLINICAL TRIAL: NCT01478126
Title: Prospective Randomized Study of Glutamin Protective Properties in Cardiac Surgery.
Brief Title: Effects of Glutamine in Ischemic Heart Disease Patients Following Cardiopulmonary Bypass
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GOP 05
Record Dates: First submitted 2011-11-16; First posted 2011-11-23 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — alanylglutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glutamine (Experimental): Intravenous glutamine infusion perioperatively and 24 hours after surgery
  Interventions: Drug: N(2)-L-Alanine L-Glutamine dipeptide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N(2)-L-Alanine L-Glutamine dipeptide — Intravenous infusion of glutamine in total dose of 2 g/kg/day (rate=2*weight/24 ml/h). Infusion starts in operating room and ends next day after the surgery.
  Other Names: Dipeptiven (N(2)-L-Alanine L-Glutamine dipeptide)
  Arms: Glutamine
Drug: Placebo — Intravenous infusion of 0,9% solution of NaCl, rate=2*weight/24. Infusion starts in operating room and ends next day after the surgery.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether perioperative glutamine administration possess protective properties on internal organs (heart and gut) in patients with coronary atherosclerosis, operated under cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with coronary artery disease operated on under cardiopulmonary bypass

Exclusion Criteria:

* Ejection fraction<40%
* Viral hepatitis
* Liver cirrhosis
* Cholecystitis
* Pancreatitis
* Chronic severe gastrointestinal disease
* Surgery on gastrointestinal tract in patient's medical history

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Troponin I | Induction to anaesthesia, 30 min after cardiopulmonary bypass, 6, 24 hours after CPB

SECONDARY OUTCOMES:
Liver Fatty Acid Binding Protein | Induction to anaesthesia (0 hour of operation), before heparin injection (1 hour of operation), 5min after aorta unclaming, 2, 6, 24 hours after CPB
  Liver fatty acid binding protein
Intestinal fatty acid binding protein | Induction to anaesthesia (0 hour of operation), before heparin injection (1 hour of operation), 5min after aorta unclaming, 2, 6, 24 hours after CPB
  Intestinal fatty acid binding protein
alpha-glutathione s-transferase | Induction to anaesthesia (0 hour of operation), before heparin injection (1 hour of operation), 5min after aorta unclaming, 2, 6, 24 hours after CPB
  alpha-glutathione s-transferase
Alanine Aminotransferase (ALT) | Induction to anaesthesia (0 hour of operation), before heparin injection (1 hour of operation), 5min after aorta unclaming, 2, 6, 24 hours after CPB
Aspartate transaminase (AST) | Induction to anaesthesia (0 hour of operation), before heparin injection (1 hour of operation), 5min after aorta unclaming, 2, 6, 24 hours after CPB
Serum HSP-70 | Induction to anaesthesia (0 hour of operation), before heparin injection (1 hour of operation), 5min after aorta unclaming, 2, 6, 24 hours after CPB
Glutathione | Induction to anaesthesia (0 hour of operation), before heparin injection (1 hour of operation), 5min after aorta unclaming, 2, 6, 24 hours after CPB
SH-groups | Induction to anaesthesia (0 hour of operation), before heparin injection (1 hour of operation), 5min after aorta unclaming, 2, 6, 24 hours after CPB

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- [Background] Lomivorotov VV, Efremov SM, Shmirev VA, Ponomarev DN, Lomivorotov VN, Karaskov AM. Glutamine is cardioprotective in patients with ischemic heart disease following cardiopulmonary bypass. Heart Surg Forum. 2011 Dec;14(6):E384-8. doi: 10.1532/HSF98.20111074. PMID 22167767